CLINICAL TRIAL: NCT00767247
Title: Analysis of Antihypertensive Treatment Efficacy
Acronym: ATACA
Status: Terminated | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Andrey Strugovshchikov, Medical Director, Astra Zeneca, Russia
Other Study IDs: NIS-CRU-ATA-2008/1
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Arterial Hypertension
Keywords: Arterial Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Male or female with arterial hypertension

SUMMARY:
Analysis of antihypertensive treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* arterial hypertension
* intake of Atacand before study enrollment

Exclusion Criteria:

* hypersensitivity to candesartan or any other ingredient of Atacand
* liver function impairment and/or cholestasis
* severe renal insufficiency (serum creatinine > 265 µmol/L)
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Analysis of antihypertensive treatment efficacy. | measurement BP: 3 visits for 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Zateyshchikov, MD, Prof, Principal Investigator — Federal State Institution of Russian President's General Management Department
Locations (13):
- Russia (13):
  - Research Site, Arhangelsk
  - Research Site, Bryansk
  - Research Site, Domodedovo
  - Research Site, Dzerzhinsk
  - Research Site, Georgiyevsk
  - Research Site, Irkutsk
  - Research Site, Kazan'
  - Research Site, Samara
  - Research Site, Severodvinsk
  - Research Site, Vidnoye
  - Research Site, Volgograd
  - Research Site, Yekaterinburg
  - Research Site, Yessentuki